CLINICAL TRIAL: NCT03472677
Title: A Phase 1b Study to Characterize the Effect of Injection Site Cooling on Pain Experienced After CNTX-4975-05 (Trans-capsaicin) Intra-articular and Capsaicin Intradermal Injections in Healthy Volunteers and Subjects With Bilateral Painful Knee Osteoarthritis
Brief Title: The Effect of Injection Site Cooling on Pain Experienced After the Administration of CNTX-4975-05 Into the Knee
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Centrexion Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CNTX-4975i-OA-101
Record Dates: First submitted 2018-03-04; First posted 2018-03-21 (Actual); Last update posted 2018-12-19 (Actual); Status verified 2018-12

CONDITIONS: Osteoarthritis, Knee
Keywords: Osteoarthritis; Knee Pain
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis | interventions — Capsaicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Cohort 1 (Experimental): A comparison of two cooling methodologies in healthy volunteers after single intra-articular (IA) injection (15 mL) of 2% lidocaine (without epinephrine).
  Interventions: Other: Ice Pack and Cooling Device; Drug: Capsaicin
- Cohort 2 (Experimental): Controlled cooling wrap versus ice pack cooling.
  Interventions: Drug: CNTX-4975-05 (trans-capsaicin); Drug: Capsaicin
- Cohort 3 (Experimental): Controlled cooling parameters will be determined after evaluation of data from prior cohorts.
  Interventions: Drug: CNTX-4975-05 (trans-capsaicin); Drug: Capsaicin
- Cohort 4 (Experimental): Controlled cooling with knee device versus no cooling (determined after evaluation of data from previous cohorts).
  Interventions: Drug: CNTX-4975-05 (trans-capsaicin); Drug: Capsaicin

INTERVENTIONS:
Other: Ice Pack and Cooling Device — A comparison of two cooling methodologies in healthy volunteers after single intra-articular (IA) injection (15 mL) of 2% lidocaine (without epinephrine).
  Arms: Cohort 1
Drug: CNTX-4975-05 (trans-capsaicin) — Controlled cooling wrap vs ice pack cooling after single IA injection of 1 mg CNTX-4975-05 in each arm after single IA (15 mL) injection of 2% lidocaine (without epinephrine).
  Arms: Cohort 2
Drug: CNTX-4975-05 (trans-capsaicin) — Controlled cooling parameters will be determined after evaluation of data from prior Cohort(s) after single IA injection (15 mL) of 2% lidocaine (without epinephrine) and single IA injection of 1 mg CNTX-4975-05.
  Arms: Cohort 3
Drug: CNTX-4975-05 (trans-capsaicin) — Controlled cooling with knee device vs no cooling (determined after evaluation of data from previous cohorts) after single IA injection (15 mL) of 2% lidocaine (without epinephrine) and single IA injection of 1 mg CNTX-4975-05.
  Arms: Cohort 4
Drug: Capsaicin — Four intradermal injections of capsaicin, two on each forearm.

SUMMARY:
A clinical study to measure the effects of injection-site cooling on pain experienced after knee injections of capsaicin in healthy subjects and in patients with knee osteoarthritis.

ELIGIBILITY:
Cohort 1 Key Inclusion Criteria:

* Subject is aged between 18 and 45 years, inclusive.
* Subjects Body Mass Index (BMI) is between 18 and 32 kg/m^2, inclusive and subject's weight is greater than or equal to 50 kg.
* Subjects must be in good health, in the opinion of the Investigator, as determined by a medical history, physical examination, clinical laboratory tests, vital signs and 12 lead electrocardiogram (ECG).

Cohort 1 Key Exclusion Criteria:

* Subject has had a clinically significant illness that has not completely resolved in the four weeks before screening.
* Subject has a history of neurological disorder which may impact the perception of pain or impairs the subject's ability to fully participate in the trial.

Cohorts 2-4 Key Inclusion Criteria:

* Subject is aged between 45 and 75 years, inclusive.
* Subject's BMI is between 18 and 32 kg/m^2, inclusive and subject's weight is greater than or equal to 50 kg.
* Subject has a diagnosis of bilateral moderate to severe painful knee OA (subjects will be required to have a score on Pain with walking in the previous 24 hours, of 4 to 9, inclusive NPRS 0-10). The condition must be chronic with a history of painful arthritis for at least 3 months prior to entry in the study.

Cohorts 2-4 Key Exclusion Criteria:

* Subject has had a clinically significant illness, other than osteoarthritis, that has not completely resolved in the four weeks before screening.
* Subject has a history of neurological disorder which may impact the perception of pain or impairs the subject's ability to fully participate in the trial.
* Subject has used analgesic medications in the 2 days prior to dosing, except for paracetamol, as needed.
* Subject has used topical medications applied to the knee for OA pain (including capsaicin, lidocaine, prescription or OTC medications) from 90 days prior to screening through to dosing.
* Subject has been injected with corticosteroids in the knee 90 days prior to screening through to dosing.
* Subject currently uses opioids for any condition other than OA knee pain (maximum dose 15 mg hydrocodone, or equivalent, per day prescribed by a physician).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-03-21 (Actual); Primary Completion 2018-07-27 (Actual); Study Completion 2018-08-03 (Actual)

PRIMARY OUTCOMES:
Numerical Pain Rating Scale (NPRS): Injection-site Pain | Days 1 and 7
  Cohorts 2-4: Change in injection-site pain following intra-articular (IA) administration of CNTX-4975-05 (trans-capsaicin) scored using NPRS on a scale of 0 to 10 with 0 corresponding to no pain and 10 corresponding to the worst pain imaginable.

SECONDARY OUTCOMES:
IA Temperature | Days 1 and 7
  Cohorts 1-4: IA temperature measurements.
Numerical Pain Rating Scale (NPRS): Procedural Pain | Days 1 and 7
  Cohort 1: Procedural pain following single intra-articular (IA) injection (15 mL) of 2% lidocaine (without epinephrine) using NPRS on a scale of 0 to 10 with 0 corresponding to no pain and 10 corresponding to the worst pain imaginable.
Numerical Pain Rating Scale (NPRS): Procedural Pain | Days 1 and 7
  Cohorts 2-4: Procedural pain following intradermal (ID) administration of the challenge agent capsaicin as a function of temperature scored using NPRS on a scale of 0 to 10 with 0 corresponding to no pain and 10 corresponding to the worst pain imaginable.
Numerical Pain Rating Scale (NPRS): Pain with Walking | Screening through Day 42
  Cohorts 2-4: Average pain with walking over the past 24 hours scored using NPRS on a scale of 0 to 10 with 0 corresponding to no pain and 10 corresponding to the worst pain imaginable.
Knee Injury and Osteoarthritis Outcome Score (KOOS) | Screening through Day 42
  Cohorts 2-4: Calculation of KOOS for each painful osteoarthritis knee on a scale of 0 to 100 with 0 representing extreme problems and 100 representing no problems.
Patient Global Impression of Change (PGIC) | Screening through Day 42
  Cohorts 2-4: Change in knee pain for each painful osteoarthritis knee scored using PGIC on a scale of 1 to 7 with 1 representing very much improved and 7 representing very much worse.
Numerical Pain Rating Scale (NPRS): Thermal Pain | Between Days 28 and 35 inclusive; and Day 42
  Cohorts 1-4: Thermal pain approximately two weeks following intradermal (ID) administration of the challenge agent capsaicin scored using NPRS on a scale of 0 to 10 with 0 corresponding to no pain and 10 corresponding to the worst pain imaginable.

CONTACTS AND LOCATIONS:
Overall Officials: Randall M. Stevens, MD, Study Chair — Centrexion Therapeutics
Locations (1):
- MAC Clinical Research, Manchester, United Kingdom